CLINICAL TRIAL: NCT05647512
Title: A Phase I/II, Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM-305 in Patients With Relapsed or Refractory Multiple Myeloma (RRMM) and Other Plasma Cell Diseases
Brief Title: Study of LM-305 in Patients With Relapsed or Refractory Multiple Myeloma (RRMM) and Other Plasma Cell Diseases
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: According to sponsor strategy
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM305-01-102
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Relapsed or Refractory Multiple Myeloma; Other Plasma Cell Diseases
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-305 Dose Escalation (Experimental): Administered intravenously
  Interventions: Drug: LM-305
- LM-305 Combination Expansion (Experimental): LM-305 Administered intravenously Dexamethasone Orally
  Interventions: Drug: LM-305; Drug: Dexamethasone

INTERVENTIONS:
Drug: LM-305 — Administered intravenously
Drug: Dexamethasone — Administered orally
  Arms: LM-305 Combination Expansion

SUMMARY:
A Phase I/II Study of LM-305 in Patients with Relapsed or Refractory Multiple Myeloma (RRMM)

DETAILED DESCRIPTION:
A Phase I/II, Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM-305 in Patients with Relapsed or Refractory Multiple Myeloma (RRMM)

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled into the study only if they meet all of the following inclusion criteria:

1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged ≥18 years old when sign the ICF, male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1。
4. Life expectancy ≥ 6 months.
5. Subjects must show appropriate organ and marrow function in laboratory examinations

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any of the following criteria:

1. A history of other malignant tumors than multiple myeloma within 3 years prior to first dosing
2. Subjects who have severe cardiovascular disease。
3. Use of any live attenuated vaccines within 28 da ys prior to 1st dosing of IMP.
4. Child-bearing potential female who have positive results in pregnancy test or are lactating.
5. Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-18 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Cycle 1 of each cohort. Duration of one cycle is 21 days
  DLT is defined as a toxicity (adverse event at least possibly related to LM305) occurring during the DLT observation period
Adverse Events (AE) and Serious Adverse Events (SAE) | From signing the informed consent form (ICF) until 28 days after end of treatment (EOT) or accept other anti-cancer therapy
  The safety profile of LM-305 will be assessed by monitoring the adverse events

SECONDARY OUTCOMES:
Area under plasma concentration vs time curve (AUC) for LM-305 | Up to finished cycle 5 (each cycle is 21 days)
  changes in AUC over time in participants with LM-305

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Principal Investigator — The First Affiliated Hospital of Soochow University